CLINICAL TRIAL: NCT04181216
Title: Comparison of Anatomically Aligned and Conventional Total Knee Arthroplasty in the Same Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Yong In, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Anatomically aligned TKRA
Record Dates: First submitted 2019-10-30; First posted 2019-11-29 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Knee Osteoarthritis; Anatomically Aligned Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anatomically aligned total knee arthroplasty prosthesis (Experimental): Total knee arthroplasty with anatomically aligned total knee arthroplasty implant (Journey II Bi-cruciate substituting total knee system, JII-BCS, Smith & Nephew)
  Interventions: Device: Anatomically aligned total knee arthroplasty implant
- Conventaional total knee arthroplasty group (Active Comparator): Total knee arthroplasty with conventional total knee arthroplasty implant (Legion total knee system, Smith & Nephew)
  Interventions: Device: Anatomically aligned total knee arthroplasty implant

INTERVENTIONS:
Device: Anatomically aligned total knee arthroplasty implant — In same patient, one total knee arthroplasty using anatomically aligned total knee arthroplasty implant Other total knee arthroplasty using conventional total knee arthroplasty implant

SUMMARY:
Total knee arthroplasty(TKA) is a successful orthopedic surgery with excellent clinical outcome and survival. However, there are concerns about patient satisfaction in previous reports, and dissatisfaction rate of 15-30% is reported in clinical outcomes(PROMs) of some studies. Therefore, for improving the patient's outcome and satisfaction after total knee arthroplasty, it is necessary to change the design of the conventional total knee arthroplsaty implant. The knee is a joint structure with several dynamic functions, and not only the skeletal structure but also the soft tissue balance plays an important role in the function of the knee joint. New implants are being developed to overcome the limitations of conventional TKA implant, including the Journey II Bi-cruciate substituting total knee system (JII-BCS; Smith & Nephew). JII-BCS implant has normal articular geometry, more anatomical femoral shape, lateral tibial convex geometry, and asymmetrical tibial plateau, anterior and posterior cams, which has been shown in experimental studies to produce nearly normal knee movement by reproducing the actual normal anatomical alignment in vivo.

The clinical results of the kinematic effects of this anatomcally aligned change are insufficient, and there is also a lack of comparative studies with conventional total knee arthroplasty implant. The purpose of this study is to compare outcomes between anatomically aligned TKA(JII-BCS) and conventional TKA(Legion total knee system, Smith & Nephew). This study is a randomized controlled study in patients undergoing total knee arthroplasty per day. Radiologic parameter, patients preference and clinical results was investigated in both knee of same patients who received TKA during minimum 2 year follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients for bilateral total knee arthroplasty
* having medicare insurance

Exclusion Criteria:

* Rheumatoid arthritis
* Other inflammatory arthritis
* Crystal-induced arthritis
* Septic arthritis
* Neuropsychiatric patients
* Previous knee operation history
* Neuropsychiatric patients
* Patients with preoperative severe limitation of motion (Flexion contracture ≥ 20, range of motion ≤ 90)
* Patients with preoperative severe defomity of knee alignment (Varus or valgus angle ≥ 15)
* Severe obese patients (BMI ≥ 40)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Western Ontario and McMaster Universities Index(WOMAC index) | Change from baseline score to score of postoperative1 year

SECONDARY OUTCOMES:
Change in Knee Society Score | Change from baseline score to score of postoperative1 year
Change in Range of Motion | Change from baseline Range of Motion at postoperative1 year